CLINICAL TRIAL: NCT00295464
Title: Randomized Trial on Efficacy and Safety of the Antenatal Rescue Course of Glucocorticoids in Threatened Premature Birth (ACG Trial)
Brief Title: Antenatal Rescue Course of Glucocorticoids in Threatened Premature Birth
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACG Trial; Betamethasone
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-02

CONDITIONS: Respiratory Distress Syndrome; Intraventricular Haemorrhage
Keywords: Antenatal glucocorticoid; Premature birth
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Drug: Betamethasone sodium phos (drug)

SUMMARY:
Administration of steroid to the mother in imminent preterm delivery is a known effective practice to decrease the risk of respiratory distress syndrome and intraventricular haemorrhage in preterm infants if given with a week of the preterm delivery. This randomized clinical trial is performed to test the possibility whether the repeat dose of steroid results in further reduction of these diseases in case the mother is in imminent preterm delivery more than a week after the first antenatal steroid treatment.

DETAILED DESCRIPTION:
RANDOMIZED TRIAL ON EFFICACY AND SAFETY OF THE ANTENATAL RESCUE COURSE OF GLUCOCORTCOID IN THREATENED PREMATURE BIRTH (ACG trial)

Introduction

Prematurity is the main cause of neonatal mortality and morbidity. Immature infants have many serious diseases such as respiratory distress syndrome (RDS), intracranial hemorrhage (ICH), chronic lung disease (CLD), necrotizing enterocolitis (NEC) and retinopathy of prematurity (ROP). Corticosteroids have the maturational effects on fetal cardiovascular, respiratory, nervous and gastrointestinal systems (1). Antenatal corticosteroids (ANC) have been widely used for prevention of RDS and other serious diseases in preterm infants since 1972's, when the controlled trial of antepartum glucocorticoid treatment was published. Administration of s of 12 mg of betamethasone given twice intramuscularly 24 hours apart has shown to be effective (2,3,4,39). Strong evidence exists for neonatal benefits from a complete course of ANC starting at 24 hours and lasting up to 7 days after treatment (2,39). Betamethasone and dexamethasone have similar biological activity and both are associated with a significant reduction in the risk of RDS, but only betamethasone with a significant decrease of the neonatal mortality. The clinical benefit had not been documented beyond 7 days after the onset of ANC therapy. (1,2)

Several randomized studies have shown that a single course of antenatal corticosteroid treatment improves the survival of preterm infants born at 24-34 weeks gestation and decreases the incidence of RDS, ICH and NEC. ANC therapy reduces the incidence of RDS by approximately 50%.(1,2) ANC treatment also reduces the need of exogenous surfactant (4). The protective effect against RDS is thought to be due to the structural maturation of the lungs, increased surfactant synthesis, improved resistance to lung injury and improved cardiovascular adaptation. Glucocorticoid speeds up the normal thinning of the gas-exchange walls with double capillary loops between the air sacs. ANC thus accelerates the structural development of the respiratory airways, but reduces the number of alveoli. Glucocorticoid increases surfactant synthesis by enhancing maturation of the surfactant- producing type II pneumocytes and stimulating the secretion of surfactant complex (1,6,7,8,9,40). Serial doses of ANC may possibly downregulate steroid receptors resulting in decreased or disordered surfactant production.(ref) ANC has not been shown to decrease the incidence of CLD at 28 days of age either in the meta-analysis or in the recent retrospective studies (2,13,14,15).

ANC treatment is associated with maturation of the cardiovascular system and normalisation of the low blood pressure in the small premature infant at birth.(ref) This influence was evident after administration of surfactant.(4) According to meta-analysis, ANC had no effect on the incidence of PDA. However in several studies, use of ANC was associated with increased spontaneous closure of PDA(2,3,4, ).

ANC decreases the incidence of ICH in preterm infants (2,3,4). Severe prematurity decreases autoregulation of the cerebral circulation and predisposes to ICH or cerebral ischemia. Glucocorticoids accelerate differentiation of neuronal cells and possibly enhance maturation of germinal matrix vessels (1,33,34). ANC therapy has been associated also with a lower incidence of periventricular leukomalacia (PVL) and cerebral palsy (CP), but these effects were not significant in Crowley's meta-analysis (2,3,4,5). In a recently published retrospective study, antenatal administration of betamethasone was associated with a decreased risk of PVL compared to antenatal dexamethasone or no treatment (17).

Betamethasone is clinically used as a mixture of betamethasone phosphate (6 mg) and betamethasone acetate (6 mg), providing a rapid exposure from the phosphate form and a sustained exposure from the acetate form. Maximal fetal serum level of betamethasone was attained 1-2 hours after ANC treatment (27). The half life of antenatally administered betamethasone is about 12 hours in fetal circulation (1,36). Decrease in the incidence of RDS is evident when ANC is administered between 24 hours and 7 days before delivery. However, the incidence of ICH is decreased even with treatment initiated less than 24 hours prior to delivery (2,3,4). According to the animal studies the short term ANC (<24 hours) improves the postnatal lung function, decreases the protein leak into the lung and alters postnatal blood pressure regulation in the premature. ANC also seems to augment the postnatal neuroendocrine and endocrine responses to hypoxic challenge (28,29,30).

According to meta-analysis there is no significant decrease in birthweight and in physical or psychological development at the age 3-12 years following a single course of ANC treatment of fetuses (2,18,19). According to follow-up studies, prenatal single course of steroid treatment is safe and enhanced survival is not associated with a higher incidence of disabilities or developmental disturbances in survivors during childhood and young adulthood (2,3,5,18,19,35). Single course of ANC treatment did not increase the risk of fetal or neonatal infections or the incidence of maternal infections (2). When administered during the subclinical chorioamnionitis, ANC treatment seem to decrease the incidence of RDS, ICH, PVL and neonatal mortality without apparent increase in neonatal sepsis (32).

However, there is concern about possible negative effect of multiple course of ANC on birthweight, head circumference and growth later in childhood. Data from numerous animal studies suggest that ANC has a negative effect on pre- and postnatal growth. Most studies deal with rodents who have a short gestation and period of growth (10,11,12,37). In animal studies multidose ANC exposure has also decreased lung growth, which seems to be irreversible and persistent into adulthood (10,11,12). Also, in several animal studies ANC exposure has shown decreased brain growth and cell proliferation, which may also be due to short duration of gestation and long duration of exposure (10,11,12,37).

There are concerns about potential suppressive effects of ANC on the fetal hypothalamus-pituitary-adrenal axis. Transient suppression of the pituitary-adrenal glands in preterm infants whose mothers have received 1-2 doses of antenatal glucocorticoid, reportedly recovers within 7 days of life (23,24,25,26,36). Infants delivered shortly after one course of ANC are normally responsive to stress after birth (e.g. RDS and asphyxia).(36)

Clinical practice administering antenatal corticosteroids varies greatly between individual centers during the late 1990's. The practice of repeating the course of ANC has become widespread. However the safety or efficacy of serial courses of glucocorticoid is not known. According to recently published non-randomized studies there is conflicting data on growth and neonatal morbidity of infants exposed to single vs. multiple course of ANC (13,14,15). There is also concern particularly in women with prolonged premature rupture of fetal membranes (PPROM) that repetitive doses may increase maternal and fetal infections (21,22). In a retrospective study the multiple course of ANC was associated with an increased incidence of maternal postpartum infections (13).

The effect of multiple courses of ANC on the HPA-axis is not well known. In recent studies a mild adrenal suppression was evident in some of the preterm infants whose mothers received more than eight courses of ANC (15). It has also been proposed that perinatal stress and exposure to corticosteroids induces long lasting changes in HPA-axis and is associated with a decrease in stress induced CRH release in adulthood (24,34). However, there is no existing data about function of HPA-axis in young adults, who have been exposed to antenatal corticosteroids during fetal life.

There is insufficient data about optimal interval of ANC administration. According to recent studies there is not additive positive effects of the practice of repeating the course of ANC at 7 days intervals. However, it is known that the positive influence of the one course of ANC is not evident after 7 days of administration. It is interesting whether one additional rescue course of ANC given within 24 hours before premature delivery is more effective than single course of ANC. No prospective studies or randomized, controlled trials comparing single versus second rescue course of antenatal corticosteroids have been published.

Specific aim and hypothesis

The present aim is to study whether in recipients of ANC a single dose of betamethasone given shortly before spontaneous or elective premature birth (gestation 24 + 0 - 33 + 6 wk) improves the neonatal outcome without causing serious side effects. According to protocol, aim is to start the placebo or the second rescue course of ANC in 48 hours before expected delivery. The first hypothesis states that administration of second rescue course of ANC is more effective than the single course of ANC in increasing the intact survival at term of all infants without major neonatal morbidity, defined by the protocol. The principal outcome is survival of premature infants without major morbidity until the age of 36+0 weeks and survival of infants born at term during early neonatal period without the major morbidity, as defined by the protocol.

Study design

Present study is a multicenter, randomized, blinded, placebo-controlled trial comparing the benefits and side effects of single vs. second rescue course of antenatal corticosteroid.

Entry criteria

The pregnant women will be eligible for the trial entry if all following criteria are met:

* administration of a course of antenatal corticosteroid at least 7 days before the trial entry
* gestational age is less than 33.0 weeks 6 days*
* very high risk of premature delivery**
* none of the following therapies complications or therapies maternal long term systemic corticosteroid therapy severe clinical chorioamnionitis (maternal fever, increased CRP or another acute phase protein, uterine tenderness) lethal disease of the fetus
* informed consent obtained
* premature rupture of membranes is not contraindication for the trial entry

  *Gestational age will be calculated from the mother's last menstrual period and confirmed by ultrasound before 20 weeks' gestation. In case the discrepancy in the estimates exceeds two weeks, ultrasound date is accepted.

  **Very high risk of premature delivery is described as follows:
* elective delivery within within 4-48 hours, as indicated by the obstetrician on the basis of the clinical status of the mother and/or the fetus
* very high risk of spontaneous delivery within 4-48 hours, i.e.
* cervix is open > 3 cm
* contractions of the uterus at 5-10 min intervals
* rupture of the membranes after the first course of ANC
* fetal and/or maternal indication for elective premature delivery or cesarean section

Trial entry

The investigator or his/her designated representative will evaluate the pregnant women for the above eligibility criteria. Administration of one course of antenatal glucocorticoid identifies the pregnant mothers that are potentially eligible to present study. Oral and written informed consent will be obtained from the women (if appropriate). The study entry (randomization and administration of the drug) takes place when all entry criteria are met. The parturient and her randomization number will be recorded on the trial data form and on patient records to enable later description of the women and to assist follow up. At the time of delivery the infants of the trial participants will be recorded to the trial data form and on patient records.

Randomization

The eligible women will be randomly and blindly assigned to receive either betamethasone or saline placebo. The randomization will take place separately in each Center according to the following strata:

I gestation at entry less than 28.0 weeks + 0 days and singleton pregnancy

II gestation at entry 28.0 weeks + 0 days or more but less than 33.0 weeks + 6 days and singleton pregnancy

III gestation at entry less than 28.0 weeks + 0 days and multiple pregnancy

IV gestation at entry 28.0 weeks + 0 days or more but less than 33.0 weeks + 6 days and multiple pregnancy

Study intervention

The first course of ANC prior to the trial entry will be given according to the clinical indications of the Center. Administration of further courses of ANC before the trial entry will disqualify the mother from the ACG trial. The study course of betamethasone or placebo will be given to each eligible woman at least 7 days after the first course of ANC. After the entry criteria are met betamethasone (12mg) or placebo (normal saline) will be drawn to a sealed syringe containing the randomization number. The drug or placebo is administered intramuscularly.

Within 1 hour the betamethasone dose increases the fetal serum levels of glucocorticoid to those obtained during neonatal stress

Other obstetric and neonatal management

Other management given to the participating women will be decided by the obstetrician. After the entry to the trial administration of ANC outside study protocol is not allowed. In an event premature delivery did not occur after ACG, any further administration of ANC is not indicated. The premature infants are treated in whatever way their condition demands, the decision is made by pediatrician. The ACG trial infants born after 33.0 + 6 weeks of pregnancy are included in the neonatal and the follow-up studies.

Fetuses that died after the trial entry will be recorded. The pathologic examination of these fetuses is strongly encouraged.

Measurement of outcome

Primary outcome of the trial:

Term birth or survival of the infants at the gestational age of 36.0 weeks + 0 days without any of the following:

RDS need of supplemental oxygen > 48 h or surfactant therapy and characteristic radiographic findings

Severe ICH (grades 3-4) infants born in term will be evaluated by ultrasound

Maternal-antenatal outcomes:

Clinical chorioamnionitis Any maternal infection Fetal death

Secondary outcomes after birth:

CLD requirement of supplemental oxygen at 36 weeks' postmenstrual age PVL (gr 3-4) Severe NEC (Bell stages 3-4) perforation of the intestine intestinal pneumatosis air in portal vein ROP according to The International Classification of Retinopathy of Prematurity

Neonatal infections early neonatal infections (onset < 72 hours) proven nosocomial bacterial or fungal sepsis during neonatal period (days 3-28) Gastrointestinal bleeding or perforation Number of days on assisted ventilation Number of days on supplemental oxygen Duration of primary hospital stay Growth characteristics at birth

Treatments requirements:

surfactant postnatal steroids indomethacin for PDA PDA surgery

Primary outcome at follow up study

Survival without neurologic, sensory or neuromotor impairment at the age 2 years, corrected for gestation. All infants will be studied. For the high-risk group, the following indices and studies will be performed:

Mental Development Index (MDI) (<70) Psychomotor development will be measured by Bayley Scale (PDI) Behavioral development index (percentile) Definition of abnormalities in neurological status, speech development, major visual handicap and hearing defect

Secondary outcomes during the follow-up:

Growth characteristics during the first two years of corrected age Recurrent infections Reactive airway disease Hospital treatment during early childhood

Data collection

Information will be collected at the time of delivery, during the hospital stay and when the baby leaves the hospital or dies. Perinatal data will include prenatal history, assessment of entry criteria and following information of postnatal condition: blood pressure monitoring, assessment of growth at birth, day 28 and at 36 weeks gestational age (height, weight and head circumference). Cranial ultrasound will be made on all infants at least between days 4-8 of life and at 36.0 w + 0 d (± 3 days) gestational age or before discharge. The worst grade of ICH and PVL will be reported. The first ophthalmologic examination for retinopathy of prematurity will be done 4 to 7 weeks after birth or at 32 weeks gestational age.

Clinical status will be assessed at the time of discharge. The cause of death will be defined when possible at autopsy.

The surviving children will be studied at two years of age (corrected for gestational age). Their growth and neurodevelopment will be evaluated using a questionnaire and a clinical evaluation.

Sample size justification

The primary goal of the study is to detect the effects of two vs. single course of ANC on survival without RDS and/or severe ICH (grade 3-4) by 36 weeks + 0 days of gestational age.

Sample size analysis is based on morbidity and mortality from the Finnish perinatal statistics (National Research and Development Centre for Welfare and Health) and from Vermont Oxford Network Database (VON). We estimate that a second additional dose of betamethasone would increase the survival without RDS and severe ICH from 50% to 62.5%. According to power analysis the sample size of 220 women would be required in each arm to reject the null hypothesis with and α of 0.05 and power of 80%.

The aim of the follow up study is to find out that one course of ANC result in equal or better neurodevelopmental outcome at the corrected age of two years, compared a single course of ANC.

Statistical analysis

Primary outcome

Analysis of the primary outcomes will be based on an intention to treat analysis of all randomized subjects. Another analysis will be performed excluding infants who had congenital lethal malformation that was not detected at the onset. The outcome will be compared for the two vs. single course of ANC using the Mantel-Haenszel chi square test stratifying by the prenatal variables.

Secondary outcomes

The frequencies of categorical outcomes will be compared using appropriate chi square tests. The growth parameters, duration of ventilation, supplemental oxygen administration and hospitalization will be compared using analysis of variance or nonparametric tests when applicable. Survival rate will be compared using chi square tests and survival to term using survival analysis.

Interim analysis

The neonatal and the follow-up results for adverse outcomes will be prepared by the Data Safety Monitoring Committee when altogether 350 study infants have reached to the term or when the trial has been going on for 24 months, whichever comes first.

Ethical considerations

A written informed consent will be obtained from all the parents of the infants before the enrollment. The participation in the study does not cause any extra cost to the mother or the family. Participation is voluntary and withdrawing from the study is possible whenever desired during the pregnancy, the hospital stay or during the follow up period. Withdrawal does not affect the treatment or the follow up of the infant or the mother. If desired, approval from the ethical committees of each participating center will be obtained.

Publication policy

The perinatal-neonatal trial and the follow up study will be published separately. The list of authors includes Antenatal Multiple Betamethasone Trial Study Group (AMBTS). Each participant of the study from each Center will be listed. Each Center has an antenatal and a postnatal trial coordinator.

Ancillary studies

The participants are free to perform ancillary studies provided that a separate protocol, submitted together with the present one, is accepted by the local ethics committees.

ELIGIBILITY:
Inclusion Criteria:

The pregnant women will be eligible for the trial entry if all following criteria are met:

* administration of a course of antenatal corticosteroid at least 7 days before the trial entry
* gestational age is less than 33.0 weeks 6 days*
* very high risk of premature delivery**
* none of the following therapies complications or therapies maternal long term systemic corticosteroid therapy severe clinical chorioamnionitis (maternal fever, increased CRP or another acute phase protein, uterine tenderness) lethal disease of the fetus
* informed consent obtained
* premature rupture of membranes is not contraindication for the trial entry

  *Gestational age will be calculated from the mother's last menstrual period and confirmed by ultrasound before 20 weeks' gestation. In case the discrepancy in the estimates exceeds two weeks, ultrasound date is accepted.

  **Very high risk of premature delivery is described as follows:
* elective delivery within within 4-48 hours, as indicated by the obstetrician on the basis of the clinical status of the mother and/or the fetus
* very high risk of spontaneous delivery within 4-48 hours, i.e.
* cervix is open > 3 cm
* contractions of the uterus at 5-10 min intervals
* rupture of the membranes after the first course of ANC
* fetal and/or maternal indication for elective premature delivery or cesarean section

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440
Dates: Start 2001-05

PRIMARY OUTCOMES:
Intact survival without RDS and/or severe (gr 3-4) ICH
Follow-up study at corrected age of two years

SECONDARY OUTCOMES:
A number of diseases in preterm infants
Number of mothers with premature delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mikko N Hallman, MD, Study Director — Children's Hospital, Univ. of Oulu; Outi M Peltoniemi, MD, Principal Investigator — Children's Hospital, Univ. of Oulu; Pentti Jouppila, MD, Study Director — Oulu Central Hospital, Dept. of Obstetrics & Gynecology
Locations (10):
- Finland (10):
  - Helsinki University Central Hospital, Finland, Helsinki
  - Joensuu Central Hospital, Joensuu
  - Jyväskylä Central Hospital, Jyväskylä
  - Kuopio University Central Hospital, Kuopio
  - Lahti Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Central Hospital of Pori, Pori
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku Central Hospital, Turku

REFERENCES:
- [Derived] Pesonen AK, Raikkonen K, Lano A, Peltoniemi O, Hallman M, Kari MA. Antenatal betamethasone and fetal growth in prematurely born children: implications for temperament traits at the age of 2 years. Pediatrics. 2009 Jan;123(1):e31-7. doi: 10.1542/peds.2008-1809. Epub 2008 Dec 15. PMID 19074961